CLINICAL TRIAL: NCT05341323
Title: Comparison Between Peri Tonsillar Infiltration of Ketamine or Bupivacaine for Post Tonsillectomy Analgesia
Brief Title: Peri Tonsillar Infiltration of Ketamine or Bupivacaine for Post Tonsillectomy Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Abdallah Abozaid, Resident doctor at otorhinolaryngiology, head and neck surgery department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Soh_Med_22_02_07
Record Dates: First submitted 2022-04-03; First posted 2022-04-22 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Post Operative Pain
Keywords: Ketamine; Bupivacaine; tonsillectomy; analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Ketamine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group K1 Ketamine (Active Comparator): pre-incisional submucosal infiltration of ketamine .5 mg/kg in the Peritonsillar area
  Interventions: Drug: Ketamine.
- Group B1 Bupivacaine (Active Comparator): pre-incisional submucosal infiltration of Bupivacaine .25 % in the Peritonsillar area
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Ketamine. — Peritonsillar infiltration of ketamine
  Arms: Group K1 Ketamine
Drug: Bupivacaine — peritonsillar infiltration of Bupivacaine
  Arms: Group B1 Bupivacaine

SUMMARY:
Comparison between the analgesic effect of local infiltration of either Bupivacaine or ketamine in the peritonsillar area before the incision of tonsillectomy to achieve postoperative analgesia

ELIGIBILITY:
Inclusion criteria

* 3-20 years old patients
* elective tonsillectomy or adenotonsillectomy with or without ventilation tube application.

Exclusion criteria

* allergy to bupivacaine or ketamine
* coagulopathy
* endocrine, neuropsychiatric or cardiopulmonary dysfunction
* increase intracranial pressure (ICP)
* psychiatric illness, history of seizure, patients under chronic analgesic treatment
* history of peritonsillar abscess, tonsillar malignancy.

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-02 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 60 minutes postoperatively
  The pain will be assessed using modiﬁed Hannallah pain scale which includes blood pressure, movement, agitation and posture where zero is the least pain and 2 is the worest necessitating rescue analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahem Risk, Professor, Study Director — Professor of ENT; Osama Elshrief, Professor, Study Chair — Dean of Faculty of Medicine
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt